CLINICAL TRIAL: NCT00078247
Title: Delaying HIV Disease Progression With Punctuated Antiretroviral Therapy in HIV-Associated Tuberculosis
Brief Title: Anti-HIV Drugs for Ugandan Patients With HIV and Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Makerere University (Other)
Responsible Party: Christopher C. Whalen, MD, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AI051219-01A2 (NIH); 1R01AI051219-01A2 (NIH)
Record Dates: First submitted 2004-02-20; First posted 2004-02-23 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Antiretroviral Therapy; Africa
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — abacavir; Lamivudine; Zidovudine

ARMS (2):
- 1 (Experimental): Participants will receive 6 months of ARV therapy and treatment for TB
  Interventions: Drug: Abacavir; Drug: Lamivudine; Drug: Zidovudine; Drug: Tuberculosis treatment
- 2 (Experimental): Participants will not receive ARV therapy until CD4 counts drop below 250 cells/mm3. All participants will receive treatment for TB.
  Interventions: Drug: Abacavir; Drug: Lamivudine; Drug: Zidovudine; Drug: Tuberculosis treatment

INTERVENTIONS:
Drug: Abacavir — 300 mg tablet taken orally twice daily
Drug: Lamivudine — 300 mg tablet taken orally daily
Drug: Zidovudine — 300 mg tablet taken orally twice daily
Drug: Tuberculosis treatment — Tuberculosis treatment

SUMMARY:
This study is designed to determine whether 6 months of anti-HIV drugs given along with tuberculosis treatment will delay the onset of AIDS in HIV infected African patients.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a common and serious complication of HIV infection in the developing world, especially in sub-Saharan Africa. Since the emergence of the HIV epidemic in Africa, the incidence rates of TB have risen dramatically, overwhelming national TB control programs across the continent. Over 50% of TB patients presenting to TB clinics in Africa are HIV infected. These patients often present in the early stages of HIV infection.

Recent World Health Organization guidelines on the management of HIV-associated pulmonary TB recommend antiretroviral (ARV) therapy in patients with CD4 cells less than 200 cells/mm3, but not for HIV infected TB patients who present with a high CD4 count. In Uganda, over half of HIV infected patients with active TB present to TB clinics with CD4 counts above 200 cells/mm3, and there is evidence that coinfected patients with a high CD4 count should be treated with ARV therapy. First, mortality in HIV-associated TB is high, even when patients respond to effective anti-tuberculosis therapy. Second, excess mortality associated with TB is most evident when CD4 counts are above 200 cell/mm3. Third, in coinfected patients, TB results in prolonged immune activation, which may enhance viral replication and accelerate the decline of CD4 cells.

This study will evaluate whether short-term ARV therapy of abacavir sulfate, lamivudine, and zidovudine given during treatment of active TB will slow progression of HIV disease in TB patients with CD4 counts of at least 350 cells/mm3. The study will also assess the possible risks (e.g., drug toxicities and resistance) and benefits (e.g., more rapid clearance of mycobacterium tuberculosis and reduced TB relapse) of punctuated ARV therapy.

Participants in this study will be HIV infected TB patients with CD4 counts of at least 350 cells/mm3. All participants will receive treatment for TB. Participants will be randomly assigned to receive 6 months of ARV therapy or to delay ARV therapy until CD4 counts drop below 250 cells/mm3. The participants will be followed for 2 years; CD4 counts will be compared between groups.

This study will also follow a group of HIV infected patients without active TB to quantify the extent to which CD4 cell decline is accelerated with active TB and to determine the extent to which a decline is neutralized in patients who receive punctuated ARV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary TB (AFB smear-positive or culture-positive)
* HIV infected
* CD4 count greater than 350 cells/mm3
* Residence within 20 km of Kampala, Uganda
* Willing to use acceptable forms of contraception during the study and for 6 weeks after stopping study medication
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Pregnancy

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2004-10

PRIMARY OUTCOMES:
CD4+ decline (slope) | Throughout study
Time to AIDS | Throughout study

SECONDARY OUTCOMES:
Safety | Throughout study
Response to antituberculous therapy | Throughout study
Immune reconstitution | Throughout study
Viral drug resistance | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Whalen, MD, Principal Investigator — Case Western Reserve University; Roy Mugerwa, MD, Principal Investigator — Makerere University; Diane Havlir, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Makerere University Medical School, Kampala, Uganda

REFERENCES:
- [Derived] Chamie G, Charlebois ED, Srikantiah P, Walusimbi-Nanteza M, Mugerwa RD, Mayanja H, Okwera A, Whalen CC, Havlir DV. Mycobacterium tuberculosis microbiologic and clinical treatment outcomes in a randomized trial of immediate versus CD4(+)-initiated antiretroviral therapy in HIV-infected adults with a high CD4(+) cell count. Clin Infect Dis. 2010 Aug 1;51(3):359-62. doi: 10.1086/654799. PMID 20569064